CLINICAL TRIAL: NCT05949814
Title: EASY-TESTS: Evaluation of the Acceptability of Pre-exposure Prophylaxis (PrEP) Among Men Who Have Sex With Men (MSM) Who Accepted Targeted HIV/STI Testing, Recruited Through a Community-based Outreach Approach, Both Digital and In-person.
Acronym: EASY-TESTS
Status: Completed | Type: Observational
Sponsor: Centre de santé sexuelle Le 190 (Other)
Collaborators: Pitié-Salpêtrière Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CSS1
Record Dates: First submitted 2023-07-10; First posted 2023-07-18 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: HIV Infections; STI
Keywords: HIV; Test; Pre-exposure prophylaxis
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HIV-negative men who have sex with men (MSM) and transgender persons
  Interventions: Diagnostic Test: acceptability of a PrEP program among HIV-negative MSM and TG

INTERVENTIONS:
Diagnostic Test: acceptability of a PrEP program among HIV-negative MSM and TG — STI screening by rapid tests and self-sampling after contact on a geolocated community application or a community physical place of sociability

SUMMARY:
Acceptability of a PrEP program among MSM and TG visiting a geolocated community application or a community physical place of sociability and having accepted a targeted screening for HIV, Hepatitis B, C and STIs.

DETAILED DESCRIPTION:
HIV infection is a transmissible infection that remains a major public health concern in 2021, with an estimated 38.4 million people living with HIV worldwide and around 2.5 million new infections. Despite therapeutic progress, wide access to screening, in France in particular, HIV infection continues to spread among the populations most exposed to this virus.

In France, 5,000 people discovered their HIV seropositivity in 2021. 44% of them are men who have sex with men (MSM), of whom more than a quarter (27%) were born abroad. 2% of new diagnoses concern transgender people2. Nearly half of people who discover their HIV status live in Paris and Île de France.

The incidence of HIV infection remains high among the key population of men who have sex with men. That of sexually transmitted infections (STIs) is increasing with more frequent screening, in particular with the introduction of HIV pre-exposure prophylaxis (PrEP). A national assessment in 2022 shows that PrEP remains mainly used by MSM, urban, educated and economically advantaged. The large number of new HIV infections each year among MSM encourages the identification of preventive actions to go to those who do not protect themselves from HIV by PrEP, do not screen themselves for STIs.

Strategies for screening and prevention of STIs and HIV must be massively encouraged and facilitated by various innovative approaches. It is important to reach out to populations who rarely see caregivers for various reasons such as social/administrative vulnerability, psychological vulnerability, non-disclosure of conditions of sexual exposure (sex workers, MSM) . The various studies show that about 40% of MSM do not report their sexual orientation to their general practitioner, and find themselves faced with a presumption of heterosexuality in the primary care system.

The 190 center is the first sexual health center created in France, in 2010. Since then, it has continued to develop expertise in Lesbian, Gay, Bisexual, Trans (LGBT+) health and, more particularly, geared towards gay health. It is one of the main centers to have implemented PrEP, as part of a range of care combining screening and treatment of STIs, specialized monitoring of HIV infection, management of the mental health of users, support for users of psychoactive products in a sexual context (Chemsex He opened THE ANTENNA in the premises of SPOT with the aim of developing innovative strategies in partnership with community guides.

The AIDES association, created in 1984, is one of the most important associations in the fight against HIV in the world, and the main one in France. It has developed many strategies, largely based on the knowledge that people most at risk/concerned by HIV-AIDS have of their communities. AIDES has opened Le SPOT in Paris, a free reception center for sexual health and harm reduction, primarily targeting an MSM population highly vulnerable to HIV infection or viral hepatitis.

Combining the activities of SPOT and L'ANTENNE makes it possible to combine the know-how of a place of community intervention and, beyond that, of the employees and volunteers of the AIDES association, with the practice of caring for a sexual health center that is today a reference in its field of expertise. The two structures focus their development on the implementation of new actions aimed at reducing the hidden epidemic of HIV infection and viral hepatitis.

The clinical research team of the Infectious Diseases department has extensive historical experience in HIV, invested in clinical research since the 1990s, and experience acquired in sexual health (PrEP, STI) with participation in studies national ANRS PREVENIR, DOXYVAC, Ganymede.

In total, taking into account the data from different studies, taking into account our respective experiences and know-how, we postulate the following hypotheses:

1. MSM and TG community dating applications and places of sociability constitute an interface of great interest for reaching an audience that does not spontaneously go to places of care adapted to their specificities in terms of health risk vis-à-vis -vis HIV and STIs.
2. The experience of the community guides, employees or volunteers, of the AIDES association makes it possible to recruit, on these applications and places, the public sought following spear-phishing strategies.
3. The screening proposal as it is designed (use of Rapid Diagnostic Orientation Tests for serological screening, bacteriological self-sampling with dematerialized rendering), responds well to a request from these users who, in fact, do not would not use mainstream offerings or places identified as offering and prescribing PrEP.
4. Through an "all-in-one" facilitated screening proposal, in a single place, free of charge, without an appointment, with immediate results, it becomes possible to bring users who would be remote, through ignorance, lack of interest, or because of negative representations of the tool or the related monitoring.

Based on a conversion rate of 3% of contacts into appointments, the objective of 24,333 contacts over one year is realistic given the difference in population density between the Center Val de Loire region (65, 7 inhabitants per km2) and the Île-de-France region (1020.8 inhabitants per km2).

This is an observational, prospective study, over 6 months, offering MSM and TG attending a geolocated community application or a community physical place of sociability, targeted screening for HIV infection, hepatitis B, C and STIs and their management in the PrEP strategy and treatment/prevention of STIs adapted to the results.

ELIGIBILITY:
Inclusion Criteria:

* Cisgender men, transgender men, and transgender women reporting sexual relations with men
* Age 18 years old
* Accepting an STIs screening after contact through a geolocated community application or a physical place of community sociability
* Given oral non-opposition to the anonymized use of the collected data

Exclusion Criteria:

* Planned stay in France <1 month
* Person under legal guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men who have sex with men (MSM) and transgender (TG) individuals
Sampling Method: Non-Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2023-07-30 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
To assess the proportion of HIV-negative participants accepting PrEP at M1 (PrEP-naive or restarting after interruption), for whom PrEP was indicated at D0 | Month 1
  The proportion of HIV-negative participants accepting PrEP at M1 (PrEP-naive or restarting after interruption), for whom PrEP was indicated at Day 0.

SECONDARY OUTCOMES:
To assess rate of acceptance of screening for STIs (HIV, Hepatitis B (HBV), Hepatitis C (HCV), syphilis) by rapid diagnostic orientation test among contacts | Day 0
  Use the Rapid diagnostic orientation test for STIs with INSTI multiplex HIV/Syphilis, + INSTI HCV + TOYO kit HBs Ag / antiHBS ab
To assess the proportion of new HIV diagnoses/known HIV-positive status | Day 0
  Use the Rapid diagnostic orientation test for HIV with INSTI multiplex HIV/Syphilis
To assess the proportion of persons with STI and type of STI (syphilis, chlamydia, gonococcus) | Day 3
  Use the Rapid diagnostic orientation test for HIV with INSTI multiplex HIV/Syphilis and by self-sampling for chlamydia and gonococcus

CONTACTS AND LOCATIONS:
Overall Officials: Michel Ohayon, Dr, Principal Investigator — Sexual Health Center 'Le 190'; Christine Katlama, Pr, Study Chair — Pitié-Salpêtrière Hospital
Locations (1):
- Le SPOT, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No